CLINICAL TRIAL: NCT07083544
Title: Comparing the Effectiveness of Sleep Hygiene Strategies Administration in Written vs Verbal Format in Track and Field Athletes: a Randomized Controlled Trial Study.
Brief Title: Sleep Hygiene Strategies Among Track and Field Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Roberto Codella, Professor, University of Milan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHS&FIDAL
Record Dates: First submitted 2025-07-07; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-06

CONDITIONS: Sleep; Athlete
Keywords: Sleep; Athletes; Actigraphy; Track and field; Sleep hygiene
MeSH Terms: conditions — Sleep Hygiene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CON (No Intervention): Partecipants do not received sleep hygiene in the second timepoint
- W-SHS (Active Comparator): An intervention group following 10 consecutive days of sleep hygiene strategies administered in a written format
  Interventions: Behavioral: Written Sleep Hygiene Strategies (W-SHS)
- V-SHS (Active Comparator): An intervention group following 10 consecutive days of sleep hygiene strategies administered in a verbal format throught an educational session
  Interventions: Behavioral: Verbal Sleep Hygiene Strategies (V-SHS)

INTERVENTIONS:
Behavioral: Written Sleep Hygiene Strategies (W-SHS) — Participants assigned to the W-SHS group received a printed handout containing general sleep hygiene strategies. These strategies were designed to improve sleep quality and included recommendations on maintaining a consistent sleep-wake schedule, minimizing light exposure before bedtime, avoiding screens and heavy meals in the evening, optimizing the sleep environment (e.g., room temperature, noise), and managing nap timing. Participants were instructed to apply these strategies consistently for 10 consecutive days. No individual guidance was provided.
  Arms: W-SHS
Behavioral: Verbal Sleep Hygiene Strategies (V-SHS) — Participants in the V-SHS group received the same general sleep hygiene strategies as the W-SHS group, but delivered through a one-on-one verbal education session. A trained researcher in sleep and sport science conducted a 40-minute session with each athlete, explaining each strategy and offering personalized clarifications and suggestions. Participants were then instructed to implement these strategies over a 10-day period.
  Arms: V-SHS

SUMMARY:
This study aims to evaluate whether different ways of delivering sleep hygiene strategies (SHS)-written materials versus one-on-one verbal instruction-affect sleep behaviors in track and field athletes. Sleep is essential for athletic recovery and performance, yet many athletes struggle to get enough rest due to both lifestyle and sport-related factors.

Sixty-six athletes were randomly assigned to one of three groups: a control group with no intervention, a group receiving SHS in written form, and a group receiving SHS through a personalized verbal session with a sleep specialist. The intervention lasted 10 consecutive days, and the same strategies were shared with both intervention groups. These strategies included advice on bedtime consistency, reducing screen use before sleep, improving sleep environment, and managing naps.

To monitor changes, participants wore an actigraphy device and completed sleep and training diaries during a 10-day baseline period (before SHS) and again during the 10-day intervention period. Researchers assessed objective sleep parameters like total sleep time, sleep efficiency, and sleep latency, as well as subjective habits using the Sleep Hygiene Index questionnaire.

DETAILED DESCRIPTION:
Sleep is vital for athletes, supporting both physical recovery and mental performance. Despite this, many athletes sleep less than recommended due to demanding training schedules, competition stress, travel, and lifestyle factors. Poor sleep impairs recovery, increases injury risk, and reduces athletic performance. One way to address this issue is through Sleep Hygiene Strategies (SHS)-a set of behavioral recommendations that help improve sleep quality and duration.

This randomized controlled trial aims to explore whether the way SHS are delivered-either through written instructions or via verbal education-affects athletes' sleep behaviors and outcomes. The study involves 66 track and field athletes, both male and female, aged 18-40, who train actively at least 2.5 hours per week. Participants are randomly assigned to one of three groups: (1) a control group with no intervention, (2) a group that receives SHS in a written format, or (3) a group that receives SHS via a 40-minute one-on-one verbal session with a trained sleep and sports science professional. The SHS are general and evidence-informed, focusing on optimizing bedtime routines, limiting electronic use before sleep, adjusting environmental factors like noise and temperature, and managing naps effectively.

Each participant has to complete a 10-day baseline sleep monitoring period and a 10-day intervention monitoring period. Sleep is measured using actigraphy (a wrist-worn movement sensor) and self-reported sleep diaries. Additional tools included a training diary and the Sleep Hygiene Index (SHI), a questionnaire is use to assess sleep-related habits.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* age between 18 and 40 years,
* FIDAL athletes,
* training for any track and field discipline for three or more times per week and over 2.5 hours of training/week.

Exclusion Criteria:

* any medical condition influencing sleep and the frequency of training in the month preceding the study,
* training or sleeping in altitude

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Total sleep time | Ten days before the administration of SHS (T0), and ten days of intervention period (T1, after the administration of SHS).
  This variable is objectively obtained by actigraphy. The total sleep time is the total amount of time a person actually spends sleeping during the night.
Sleep Latency | Ten days before the administration of SHS (T0), and ten days of intervention period (T1, after the administration of SHS).
  This variable is objectively obtained by actigraphy. The amount of time it takes to fall asleep after going to bed.
Sleep Efficiency | Ten days before the administration of SHS (T0), and ten days of intervention period (T1, after the administration of SHS).
  This variable is objectively obtained by actigraphy. The percentage of time spent asleep while in bed, calculated as TST divided by time in bed.
Wake after sleep onset | Ten days before the administration of SHS (T0), and ten days of intervention period (T1, after the administration of SHS).
  This variable is objectively obtained by actigraphy. The total duration of wakefulness occurring after initial sleep onset.
Bedtime | Ten days before the administration of SHS (T0), and ten days of intervention period (T1, after the administration of SHS).
  This variable is objectively obtained by actigraphy. The time a person gets into bed with the intention of going to sleep.
Wake up time | Ten days before the administration of SHS (T0), and ten days of intervention period (T1, after the administration of SHS).
  This variable is objectively obtained by actigraphy. The time a person finally gets out of bed to start their day.
Sleep regularity index | Ten days before the administration of SHS (T0), and ten days of intervention period (T1, after the administration of SHS).
  This variable is objectively obtained by actigraphy. A measure of how consistent sleep and wake times are from day to day.

SECONDARY OUTCOMES:
Number of training | Ten days before the administration of SHS (T0), and ten days of intervention period (T1, after the administration of SHS).
  The total count of distinct workouts an athlete completes in a week.
Weekly Training Hours | Ten days before the administration of SHS (T0), and ten days of intervention period (T1, after the administration of SHS).
  The cumulative amount of time spent exercising or training over the course of a week.
Training load | Ten days before the administration of SHS (T0), and ten days of intervention period (T1, after the administration of SHS).
  A measure that combines the intensity and duration of training to reflect the overall physical demand placed on the body.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Biomedical Sciences for Health | Università degli Studi di Milano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sargent C, Lastella M, Halson SL, Roach GD. How Much Sleep Does an Elite Athlete Need? Int J Sports Physiol Perform. 2021 Dec 1;16(12):1746-1757. doi: 10.1123/ijspp.2020-0896. Epub 2021 May 21. PMID 34021090
- [Background] Walsh NP, Halson SL, Sargent C, Roach GD, Nedelec M, Gupta L, Leeder J, Fullagar HH, Coutts AJ, Edwards BJ, Pullinger SA, Robertson CM, Burniston JG, Lastella M, Le Meur Y, Hausswirth C, Bender AM, Grandner MA, Samuels CH. Sleep and the athlete: narrative review and 2021 expert consensus recommendations. Br J Sports Med. 2020 Nov 3:bjsports-2020-102025. doi: 10.1136/bjsports-2020-102025. Online ahead of print. PMID 33144349
- [Background] Vitale JA, Borghi S, Piacentini MF, Banfi G, La Torre A. To Sleep Dreaming Medals: Sleep Characteristics, Napping Behavior, and Sleep-Hygiene Strategies in Elite Track-and-Field Athletes Facing the Olympic Games of Tokyo 2021. Int J Sports Physiol Perform. 2023 Sep 20;18(12):1412-1419. doi: 10.1123/ijspp.2023-0144. Print 2023 Dec 1. PMID 37730209